CLINICAL TRIAL: NCT02646007
Title: Autologous Bone Marrow Derived Mesenchymal Stromal Cells Transplantation for Human Avascular Necrosis of the Lunate Bone of the Wrist (Kienbock's Disease)
Brief Title: Autologous Bone Marrow Derived Mesenchymal Stromal Cells Transplantation(BM-MSC) for Kienbock's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Bone-014
Record Dates: First submitted 2015-12-03; First posted 2016-01-05 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Kienböck's Disease
Keywords: Autologous Cell therapy Kienböck's disease; bone marrow derived mesenchymal stromal/stem cell
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BM-MSC (Experimental): Bone marrow derived mesenchymal stromal/stem cells injection during decompressive surgery in patients with Kienböck's disease.
  Interventions: Biological: BM-MSC transplantation

INTERVENTIONS:
Biological: BM-MSC transplantation — Transplantation of bone marrow derived mesenchymal stem/ stromal cells in combination with bone decompression surgery in Kienböck's disease.

SUMMARY:
Kienböck's disease is characterized by avascular necrosis of the lunate wrist bone, which is usually progressive without treatment.

Cell therapy is useful in treatment of degenerated bone and mesenchymal stromal/stem cells are the best candidates for this kind of treatment.

This study examined lunate core decompression in combination with implantation of autologous bone marrow derived mesenchymal stromal cells for Its treatment potential.

Bone decompression in combination with implantation of autologous bone marrow derived mesenchymal stromal/stem cell will be done in 30 patients with Kienböck disease.

The patients will be followed at 2weeks, 3months, 6m and 12 months after implantation.

The Spss(v16) software will be used for data analysis.

DETAILED DESCRIPTION:
Kienböck's disease is characterized by avascular necrosis of the lunate wrist There is probably no single cause of avascular necrosis of the lunate. Its origin may involve multiple factors, such as the blood supply (arteries), the blood drainage (veins), and skeletal variations.

Current treatments are: at the early phase only observation. In the more advanced phases surgical techniques such as bone decompression.

A potential therapeutic strategy would be cell therapy, A source of such cells with a regenerative potential could be mesenchymal stem cells (MSCs).

The investigators will evaluate safety and efficacy of implantation of autologous BM-MSC (bone marrow-derived mesenchymal stromal cell) in 30 patients with Kienböck's disease in combination with bone decompression surgery. These patients will be followed up and data will be analyzed with spss(v16).

ELIGIBILITY:
Inclusion Criteria:

* Kienböck's disease without response to conservative treatment (physical and medical) for over 6 months
* Both genders
* Visual Analogue Scale of 4 or higher
* Hematological and biochemical analysis with no significant alterations that contraindicates intervention
* The patient is able to understand the nature of the study
* Informed written consent of the patient

Exclusion Criteria:

* Age over 65 or under 18 or legally dependent
* Infection signs or positive serology for HIV, hepatitis and syphilis
* Allergy to gentamicin, or to bovine, cattle or horse serum
* Pregnancy or lactating
* Pregnancy or breast-feeding
* Neoplasia
* Immunosuppression
* Participation in another clinical trial or treatment with another investigational product within 30 days prior to inclusion in the study
* Other conditions that may, according to medical criteria, discourage participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 3months
  The pain reduction at least 3 months after BM-MSC transplantation cells in combination with bone decompression.
Bone density | 3 months
  The improvement of bone density at least 3months after BM-MSC transplantation in MRI.

SECONDARY OUTCOMES:
Quality of life evaluated by Visual Analogue Score (VAS) | 3 months
  Improvement of quality of life inpatients after at least 3months of BM-MSC transplantation that is evaluated by Visual Analogue Score (VAS). The patients depends on their severity of the pain during daily activity choose a score between 1-10. The score will be saved in score sheets.
Infection: Presence of any sign or symptoms of infection | 1week
  presence of any sign or symptoms of infection in site of surgery during 1 week.
Cyst formation: Presence of any cyst or mass formation | 3months
  presence of any cyst or mass formation at least 3 months after BM-MSC transplantation with surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of department of Regenerative Medicine & Cell therapy center, Royan Institute; Hamidreza Mehrpour, MD, Study Director — Tehran university of medical science, department of orthopedic surgery; Mohsen Emadedin, MD, Principal Investigator — Department of Regenerative Biomedicine at the Cell Science Research Center, Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran.; Narges Labibzadeh, MD, Principal Investigator — Department of Regenerative Biomedicine at the Cell Science Research Center, Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran.
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Sadri B, Labibzadeh N, Mirmorsali L, Ebrahimi M, Bagherifard A, Arab L, Aghdami N, Madani H, Beheshti Maal A, Karimi S, Mehrpour SR, Emadedin M, Vosough M. Local Transplantation of Mesenchymal Stromal Cells Is Safe and Could Alleviate Kienbock Disease's Complications: A Clinical Trial Study. Cell J. 2024 Sep 11;26(7):446-453. doi: 10.22074/cellj.2024.2028891.1572. PMID 39290122
- See also: Related Info — http://royaninstitute.org